CLINICAL TRIAL: NCT01979497
Title: Adhesive Strips in Dermatologic Surgery: Is Cosmetic Appearance Improved?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 451808; 451808 (Other: University of California, Davis)
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Subjects Undergoing Surgical Procedure of the Skin
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture with Adhesive Stripping (Active Comparator): Buried dissolving subcuticular sutures are sued for both sides of the wound to approximate wound edges and then steri-strips for the adhesive stripped half of the scar is applied.
  Interventions: Procedure: Suture with Adhesive Stripping; Procedure: Suture without Adhesive Stripping
- Suture without Adhesive Stripping (Active Comparator): Buried dissolving subcuticular sutures are sued for both sides of the wound to approximate wound edges and then no closure material for the half of the scar is applied.
  Interventions: Procedure: Suture with Adhesive Stripping; Procedure: Suture without Adhesive Stripping

INTERVENTIONS:
Procedure: Suture with Adhesive Stripping
Procedure: Suture without Adhesive Stripping

SUMMARY:
To determine whether the addition of adhesive stripping to a wound closed with dermal sutures improves outcome of wound closure. We hypothesize that the combination of adhesive strips to a wound closed with dermal sutures does not add significant cosmetic improvement of the resultant scar.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Willing to return for follow up visit

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Unwilling to return for follow up
* Wounds less than 3 cm in length
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers 17 and under)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Split-Scar Comparison | 3 months
  Split-scar comparison of half of the wound closed with buried subcuticular sutures and overlying adhesive strips and half the wound closed with buried subcuticular sutures alone.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Derived] Custis T, Armstrong AW, King TH, Sharon VR, Eisen DB. Effect of Adhesive Strips and Dermal Sutures vs Dermal Sutures Only on Wound Closure: A Randomized Clinical Trial. JAMA Dermatol. 2015 Aug;151(8):862-7. doi: 10.1001/jamadermatol.2015.0174. PMID 25875131
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical